CLINICAL TRIAL: NCT03910842
Title: Adoptive Immunotherapy for Children CD19+ Leukemia and Non-Hodgkin Lymphoma With CD19-TriCAR-T/SILK Cell
Brief Title: Treatment of Children CD19+ Leukemia and Non-Hodgkin Lymphoma With CD19-TriCAR-T/SILK Cell Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2018-14
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-03

CONDITIONS: Non-Hodgkin Lymphoma of Intestine; Leukemia
Keywords: Non-Hodgkin Lymphoma; Leukemia; children; CD19; CAR-T; TriCAR-T; TriCAR-SILK
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-TriCAR-T/NK（SILK） (Experimental): CD19-TriCAR-T/SILK cells will be administered intravenously
  Interventions: Biological: CD19-TriCAR-T/SILK

INTERVENTIONS:
Biological: CD19-TriCAR-T/SILK — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide may be administered, followed by a single infusion of CD19-TriCAR-T cells or 4 repeat infusions of CD19-TriCAR-SILK cells.

SUMMARY:
This is a single arm, open-label, early phase Ⅰ study, to determine the safety and efficacy of CD19-TriCAR-T and CD19-TriCAR-SILK cell therapy in Children CD19+ Leukemia Non-Hodgkin lymphoma treatment.

DETAILED DESCRIPTION:
CD19-TriCAR contains an anti-CD19 scFv, a PD-L1 blocker, and a cytokine complex, enabling the CD19-TriCAR-T/SILK to simultaneously targeting the CD19 positive Leukemia or Non-Hodgkin lymphoma，blocking the inhibitory PD-L1 signal and stimulating innate T/NK cell activation and expansion, thus make it a tri- functional CAR (Tri-CAR). CD19-TriCAR-T is an autologous tri-functional CAR-T cell therapy, CD19-TriCAR-SILK is an Allogeneic tri-functional CAR- NK cell therapy, patients ineligible for leukapheresis or CAR-T therapy will be recommended for CD19-TriCAR-SILK therapy.

ELIGIBILITY:
Inclusion Criteria:

For children CD19 positive B cell leukemia：

1. All subjects must personally sign and date the Informed Consent before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. CD19-positive B-cell leukemia with histology or cytology confirmed recurrence after treatment; or progression during treatment; or after first line treatment getting a MRD negative, 2 times of MRD show>0.01% but without bone marrow morphology recurrence;
4. At least one measurable lesion;
5. Aged <18 years; or diagnosised at the age of less than 18 and relapsed within three years， determined by the investigator;
6. Expected survival ≥12 weeks;
7. Eastern cooperative oncology group(ECOG) performance status of≤2;
8. Before CD19-TriCAR-T/SILK cell infusion, systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
9. All other treatment induced adverse events must have been resolved to ≤grade 1;

For children CD19 positive B cell lymphoma：

1. All subjects must personally sign and date the Informed Consent before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. CD19-positive B-cell lymphoma with histology or cytology confirmed recurrence after treatment，defined as one or more of the following: disease progression during standard therapy；recurrence after termination of treatment；relapse after autologous hematopoietic stem cell transplantation；not suitable for stem cell transplantation or abandon stem cell transplantation due to conditional restrictions;
4. At least one measurable lesion;
5. Aged <18 years; or diagnosised at the age of less than 18 and relapsed within three years， determined by the investigator;
6. Expected survival ≥12 weeks;
7. Eastern cooperative oncology group(ECOG) performance status of≤2;
8. Before CD19-TriCAR-T/SILK cell infusion, systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
9. All other treatment induced adverse events must have been resolved to ≤grade 1;

Exclusion Criteria:

1. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring iv antimicrobials for management. (Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment);
2. Patients with symptomatic central nervous system metastasis, intracranial metastasis, and cancer cells found in cerebrospinal fluid are not recommended to participate in this study. Symptom free or post-treatment stable disease or disappearance of lesions should not be excluded. The specific selection is ultimately determined by the investigator;
3. Lactating women or women of childbearing age who plan to conceive during the time period;
4. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
5. Known history of infection with HIV;
6. Subjects need systematic usage of corticosteroid;
7. Subjects need systematic usage of immunosuppressive drug;
8. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
9. Other reasons the investigator consider the patient may not be suitable for the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
safty (Incidence of treatment-related adverse events as assessed by CTCAE v4.03) | 24 monthes
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Complete response rate[CR] (Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 24 monthes
  Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma

OTHER OUTCOMES:
Partial response rate [PR] （Partial response rate per the revised International Working Group (IWG) Response Criteria） | 24 monthes
  Partial response rate per the revised International Working Group (IWG) Response Criteria
Duration of Response （The time from response to relapse or progression） | 24 monthes
  The time from response to relapse or progression
Progression Free Survival （The time from the first day of treatment to the date on which disease progresses） | 24 monthes
  The time from the first day of treatment to the date on which disease progresses
Overall Survival （The number of patient alive, with or without signs of cancer） | 24 monthes
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Xiangling He, Principal Investigator — Hunan Provincial People's Hospital
Locations (1):
- Hunan Provincial People's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No